CLINICAL TRIAL: NCT04872868
Title: Evaluation of the Long-term Effect of a 3-month Supplementation With Holo-BLG (Food for Special Medical Purposes) in People With Allergic Rhinoconjunctivitis Caused by House Dust Mites During Inhalation Exposure to Mite Allergen in an Exposure Chamber.
Brief Title: Long-term Effect of a 3-month Supplementation With Holo-BLG on House Dust Mite Induced Allergic Rhinoconjunctivitis
Status: Completed | Type: Observational
Sponsor: Ecarf Institute GmbH (Other)
Collaborators: Bencard Allergie GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 014-P-21
Record Dates: First submitted 2021-04-23; First posted 2021-05-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-04

CONDITIONS: Dust Mite Allergy; Allergic Rhinitis
MeSH Terms: conditions — Dust Mite Allergy; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate the long-term effect of a lozenge containing beta-lactoglobulin (BLG), iron, retinoic acid, zinc and polyphenols (holo-BLG) in people with allergic rhinoconjunctivitis caused by house dust mites and the associated symptoms (symptom type and severity) during exposure to house dust mites in an Allergen Exposure Chamber (AEC).

In particular, the study aims to evaluate whether the improvements in symptoms of house dust mite-induced rhinoconjunctivitis observed after 3 months of supplementation with holo-BLG can still be detected 7 to 8 months after the last intake.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the predecessor study including complete intake of the holo-BLG lozenge for 3 months; inclusion in the final analysis set of the predecessor study
* patients with allergic rhinoconjunctivitis caused by house dust mites of any gender, aged 18-65 years
* Verbal and written informed consent

Exclusion Criteria:

* Persons <18 years
* lack of verbal and written consent
* persons who do not speak German
* seriously ill persons
* Persons with immunosuppressive medication such as systemic corticosteroids, cyclosporine
* Pregnancy and breastfeeding
* psychiatric illness
* Persons who have received or have started sublingual or subcutaneous immunotherapy (SLIT/SCIT) against house dust mites in the last 2 years before screening
* Contraindications and/or history of adrenaline intolerance and/or emergency medication.
* Concurrent use of anti-allergic medications and/or inadequate washout period of these anti-allergic medications prior to the selection process and exposure in the exposure chamber
* Use of an investigational drug 30 days/5 half-lives of the drug (whichever is longer) prior to screening
* Use of certain drugs prior to V5: Systemic corticosteroids within 3 weeks; Topical nasal corticosteroids within 2 weeks; Chromones within 7 days; Antihistamines within 72h; Antibiotics within 3 months; Pro-, Pre- and Synbiotics 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study participants must have been participated in the in the predecessor study (supplementation phase with holo-BLG) including complete intake of the holo-BLG lozenge for 3 months and must have been included in the final analysis set of the predecessor study
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
TNSS | After 120 minutes of allergen challenge
  Total Nasal Symptom Score (TNSS) in response to HDM exposure in an AEC at V1 (baseline AEC exposure) versus V5 (follow-up AEC exposure). The TNSS is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TNSS of 12.

SECONDARY OUTCOMES:
TSS | Up to 120 minutes following allergen challenge
  Total Symptom Score in response to HDM exposure in an AEC at V1 (baseline AEC exposure) versus V5 (follow-up AEC exposure). The TSS is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose), 3 eye symptoms (itchy eyes, watery eyes, and gritty feeling), 4 bronchial symptoms (wheezing, cough, breathlessness, and asthma), and 2 other symptoms (itchy palate, and itchy skin) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TSS of 39.
TESS | Up to 120 minutes following allergen challenge
  The Total Eye Symptom Score (TESS) is the sum of 3 eye symptoms (itchy eyes, watery eyes, and gritty feeling) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TESS of 9.
TBSS | Up to 120 minutes following allergen challenge
  The Total Bronchial Symptom Score (TBSS) is the sum of 4 bronchial symptoms (wheezing, cough, breathlessness, and asthma) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TBSS of 12.
VAS | Recorded at time zero (0) and every 30 minutes during exposure until 120 minutes
  Visual Analogue Scale: Before, every 30 minutes during and after the exposure patients grade the question on their well-being by putting a vertical line on a 10 cm line representing severity from 0 cm "very good" to 10 cm "very bad".
PNIF | Recorded at time zero (0) and every 30 minutes during allergen exposure up to 120 minutes
  PNIF (peak nasal inspiration flow) liter/minute.
PEF | Recorded at time zero (0) and every 30 minutes during allergen exposure up to 120 minutes
  PEF (peak expiratory flow) liter/minute.
FEV1 | Recorded at time zero (0) and 120 minutes
  Forced expiratory volume in 1 second, before and after the exposure.
FEV1/FVC | Recorded at time zero (0) and 120 minutes
  Forced expiratory volume in 1 second/forced vital capacity ratio, before and after the exposure.
rescue medication and/or emergency treatment | during and up to 24 hours after AEC exposure
  Need for rescue medication and/or emergency treatment
Adverse events with regards to the allergen exposure | up to 24 hours after AEC exposure
  Number of events and number of patients recording late-phase reactions and/or adverse events with regards to the allergen exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Becker, Study Director — Ecarf Institute GmbH
Locations (1):
- ECARF Institute GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergmann, KC., Raab, J., Krause, L. et al. Long-term benefits of targeted micronutrition with the holoBLG lozenge in house dust mite allergic patients. Allergo J Int (2022). https://doi.org/10.1007/s40629-021-00197-z